CLINICAL TRIAL: NCT03711305
Title: Randomized, Double-blinded, Placebo Controlled, Multicenter, Phase III Study of Carboplatin Plus Etoposide With or Without SHR-1316 in Participants With Untreated Extensive-Stage (ES) Small Cell Lung Cancer (SCLC)
Brief Title: Study of Carboplatin Plus Etoposide With or Without SHR-1316 in Participants With Untreated Extensive-Stage (ES) Small Cell Lung Cancer (SCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1316-III-301
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHR-1316 + carboplatin + etoposide (Experimental): Participants will receive SHR-1316 intravenously in combination with carboplatin and etoposide during the induction phase (Cycles 1-4 or 6). Thereafter, participants will receive maintenance (after induction phase) SHR-1316 until persistent radiographic PD, intolerable toxicity or withdrawal of consent.
  Interventions: Drug: SHR-1316; Drug: Carboplatin; Drug: Etoposide
- Placebo + carboplatin + etoposide (Active Comparator): Participants will receive placebo intravenously in combination with carboplatin and etoposide during the induction phase (Cycles 1-4 or 6). Thereafter, participants will receive maintenance (after induction phase) placebo until persistent radiographic PD, intolerable toxicity or withdrawal of consent.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Placebo

INTERVENTIONS:
Drug: SHR-1316 — SHR-1316 intravenous infusion will be administered during the induction phase (Cycles 1-4 or 6) and maintenance phase.
  Arms: SHR-1316 + carboplatin + etoposide
Drug: Carboplatin — Carboplatin intravenous infusion will be administered during the induction phase (Cycles 1-4 or 6).
Drug: Etoposide — Etoposide intravenous infusion will be administered during the induction phase (Cycles 1-4 or 6).
Drug: Placebo — Placebo intravenous infusion will be administered during the induction phase (Cycles 1-4 or 6) and maintenance phase.
  Arms: Placebo + carboplatin + etoposide

SUMMARY:
This randomized, double-blinded, placebo-controlled phase III, multicenter study is designed to evaluate the safety and efficacy of SHR-1316 in combination with carboplatin plus (+) etoposide compared with treatment with placebo + carboplatin + etoposide in chemotherapy-naive participants with ES-SCLC.

DETAILED DESCRIPTION:
Participants will be randomized in a 1:1 ratio to receive either SHR-1316 + carboplatin + etoposide or placebo + carboplatin + etoposide for 4-6 cycles in the induction phase followed by maintenance with SHR-1316 or placebo until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Treatment can be continued until persistent radiographic PD or or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and <= 75 years
* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system)
* Eastern Cooperative Oncology Group performance status of 0 or 1
* No prior systemic treatment or immune checkpoint inhibitor treatment for ES-SCLC
* At least 6 months treatment-free period since last chemo/radiotherapy with curative intent for limited-stage SCLC
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function
* Patients must submit a pre-treatment tumor tissue sample during the study.
* Signed inform consent form

Exclusion Criteria:• Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation

* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 1 week prior to randomization
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Malignancies other than SCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* History of autoimmune disease, including but not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease
* Prior treatment with immune checkpoint blockade therapies
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid are permitted in the absence of active autoimmune disease.
* Significant cardiovascular disease
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Treatment with systemic immunosuppressive medications within 2 weeks prior to randomization
* History of hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, carboplatin or etoposide
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Duration of Overall Survival (OS) | up to approximately 31 months
  Baseline until death from any cause

SECONDARY OUTCOMES:
Duration of Progression-Free Survival (PFS) as Assessed Using RECIST v1.1 | up to approximately 6 months
Percentage of Participants With Objective Response (OR) as Assessed by the Investigator Using RECIST v1.1 | up to approximately 31 months
  Baseline until partial response (PR) or complete response (CR), whichever occurs first
Duration of Response (DOR) as Assessed by the Investigator Using RECIST v1.1 | up to approximately 31 months
  First occurrence of PR or CR until PD or death, whichever occurs first
Percentage of Participants Alive and Without PD, as Assessed by the Investigator Using RECIST v1.1, at 6 Months and 1 Year | 6 months, 1 year
Percentage of Participants Alive at 1 Year and 2 Years | 1 year, 2 years
Percentage of Participants with Adverse Events Or Serious Adverse Events. | up to approximately 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Jilin Cancer Hospital, Jilin, Changchun

REFERENCES:
- [Derived] Long Y, Wang H, Xie X, Li J, Xu Y, Zhou Y. Updated cost-effectiveness analysis of adebrelimab plus chemotherapy for extensive-stage small cell lung cancer in China. BMJ Open. 2024 Apr 5;14(4):e077090. doi: 10.1136/bmjopen-2023-077090. PMID 38582540
- [Derived] Wang J, Zhou C, Yao W, Wang Q, Min X, Chen G, Xu X, Li X, Xu F, Fang Y, Yang R, Yu G, Gong Y, Zhao J, Fan Y, Liu Q, Cao L, Yao Y, Liu Y, Li X, Wu J, He Z, Lu K, Jiang L, Hu C, Zhao W, Zhang B, Shi W, Zhang X, Cheng Y; CAPSTONE-1 Study Group. Adebrelimab or placebo plus carboplatin and etoposide as first-line treatment for extensive-stage small-cell lung cancer (CAPSTONE-1): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Jun;23(6):739-747. doi: 10.1016/S1470-2045(22)00224-8. Epub 2022 May 13. PMID 35576956